CLINICAL TRIAL: NCT06543810
Title: Parkinson's Improvement Activated by Hula Understanding
Acronym: PAHU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSP #24723
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Pilot feasibility study for Hula intervention in PD patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hula Pilot Intervention (Experimental): Hula pilot 3 month program for PD patients.
  Interventions: Other: Hula for Parkinson's

INTERVENTIONS:
Other: Hula for Parkinson's — A feasibility study for a Hula program for Parkinson's Disease patients.

SUMMARY:
Parkinson's improvement Activated by Hula Understanding (PAHU), a pilot study, will evaluate the feasibility of hula program on patients with Parkinson's disease (PD). Hula combines several aspects-moderate physical activity, cardiovascular risk reduction, social support opportunities, and other stress-reducing qualities that have potential to prevent further neurodegeneration, improve balance and mobility, help non-motor symptoms and quality of life of PD patients in a sustainable and relatable fashion. The investigators will create a hula program specifically to the needs of patients with PD with mobility difficulty as a non-pharmacological intervention and conduct a pilot study to test the feasibility of such program. The investigators will learn from leaders of the Dance for PD (NYC), an internationally acclaimed program offering a range of dance classes for PD patients), as well as other key informants. The investigators will create once a week hula program for 3 months for PD patients and assess the feasibility of such program. Participants will undergo motor testing before and after the hula program, and will be interviewed for their feedback.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is the second most common progressive neurodegenerative disorder (after Alzheimer's disease) that is characterized by both motor and non-motor manifestations that leads to significant disability, morbidity, and mortality. The risk of PD increases with age with a prevalence of approximately 1-2% of the population over 65-years-old. The economical, physical and psychological burden of PD on patients, caregivers, families and society is enormous. Currently, there is no cure for PD. Available treatments for PD (e.g., medication and surgery) are focused on symptom control and do not fully address certain motor symptoms such as balance and voice, or non-motor symptoms such as apathy, depression and anxiety. Identification of effective treatments that addresses balance and voice, as well as non-motor symptoms, quality of life and wellbeing, is an unmet need for PD patients. Recent research has shown that exercise, including dance, can have positive effects on gait, speed, strength, balance, and quality of life for individuals with PD. However, less is known regarding how to translate and implement these promising results from short term non-pharmacological intervention into the lifestyle of patients suffering a chronic disease with mobility and cognitive difficulty. Hula, the traditional dance of Native Hawaiians and a hallmark of Hawaiian culture, has a potential to be a culturally aligned, relatable and sustainable intervention for PD patients in Hawai'i. Hula may even have broader potential for all PD patients.

Parkinson's improvement Activated by Hula Understanding (PAHU), will evaluate the impact of hula on patients with PD. Previous studies done in Hawai'i have shown hula to be an effective and meaningful non-pharmacological intervention for patients with cardiovascular disease, with improvements in physical functioning and HRQOL. Increasing evidence suggests that cardiovascular burden can either add to the brain health comorbidity, and/or have a synergistic effect on neurodegeneration. Reduction of cardiovascular risk may contribute to improved health outcomes in PD patients. Thus, hula combines several aspects-moderate physical activity, cardiovascular risk reduction, social support opportunities, and other stress-reducing qualities that have potential to prevent further neurodegeneration, improve balance and mobility, help non-motor symptoms and quality of life of PD patients in a sustainable and relatable fashion. The investigators will create a hula program specifically tailored to the needs of PD patients with mobility difficulty as a non-pharmacological intervention. To do this, investigators will learn from leaders of the Dance for PD, which was launched in NYC in 2001 and is now an internationally acclaimed program offering a range of dance classes for PD patients, and incorporate their methodology into our hula intervention. The investigators will build on prior work in Hawaii and ensure that the hula program integrated the cultural and conceptual 'heart' of hula by interviewing other key informants. In this pilot, the investigators will evaluate the feasibility, safety, resource needs and effectiveness of the 3-month hula intervention in a pilot study for people with mild to moderate PD. This pilot study will be a prospective single arm cohort study with no control group. The hula classes will be delivered in a group setting, for one (1) hour, once a week for 3 months (12 total classes). Participants will undergo motor testing before and after the hula program, and will be interviewed for their feedback.

ELIGIBILITY:
Inclusion Criteria

* Primary diagnosis of idiopathic PD confirmed by a movement disorder specialist.
* Age over 25-years-old.
* Ability to give informed consent

Exclusion Criteria:

* Presence of physical or mental health co-morbid conditions severe enough to prevent participation.
* Drug or alcohol dependence that might interfere with safe participation, based on opinion of the Principal Investigator
* Inability to attend in-person hula classes and study visits at Queens Medical Center.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Retention | 3 months
  number of participants completing final assessments/number of participants consented

SECONDARY OUTCOMES:
UPDRS-III | Baseline and 3-month follow up
  Unified Parkinson's Disease Rating Scale Part III. Multiple questions with a scale from 0-4 or 0-1, lower indicates lower symptom severity.
PDQ-39 | Baseline and 3-month follow up
  Parkinson's Disease Questionaire. 39 questions, each on a scale from 0-4. Lower values indicate reduced severity of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No